CLINICAL TRIAL: NCT02363699
Title: Effect of Endovenous Lidocaine on Analgesia and Serum Cytokines Concentration: Randomized and Double-blind Trial
Brief Title: Endovenous Lidocaine and Serum Cytokines Concentration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Collaborators: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Juliano Ferreira, PhD, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIDOCAINE X CYTOCINES
Record Dates: First submitted 2015-02-04; First posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Cholelithiasis
Keywords: cholelithiasis; Cytokines; under general anesthesia
MeSH Terms: conditions — Cholelithiasis | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Active Comparator): Group treated with lidocaine solution
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Group treated with saline solution
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Lidocaine — Lidocaine was administered in bolus of 1.5 mg.kg-1 at the start of the procedure and maintained at a dose of 3 mg.kg-1.h-1 until one hour after the end of the procedure. Solution of 0,3% lidocaine was used, so that the infusion rate was equal to the weight of the patient.
  Other Names: Xilocayne; Lidocaine hydrochloride
  Arms: Lidocaine
Drug: Saline solution — Saline solution was administered in bolus of 1.5 mg.kg-1 at the start of the procedure and maintained at a dose of 3 mg.kg-1.h-1 until one hour after the end of the procedure.
  Arms: Placebo

SUMMARY:
Ineffective treatment of postoperative pain may cause organic damage and chronic pain. Nevertheless, opioids, the leading drugs used for this purpose, present side effects that sometimes restrict their usability. In a multimodal context, new postoperative analgesia techniques have been developed focusing in the reduction of opioid use and their adverse effects, as well as postoperative chronic pain prevention. In this background, continuous intravenous infusion of lidocaine during perioperative period has shown to be promising. This trial aimed to compare postoperative analgesia, opioid consumption, duration of ileus and length of hospital stay and IL-1, IL-6, IL-10, α TNF and γ IFN levels in patients undergoing to laparoscopic cholecystectomies who received intravenous lidocaine in comparison to a control group. Intravenous lidocaine in the perioperative period of laparoscopic cholecystectomies was not able to reduce postoperative pain, opioid consumption, and duration of ileus or length of hospital stay. However, its anti-inflammatory effect was evidenced by the significant changes in the studied cytokines.

DETAILED DESCRIPTION:
Forty-four patients undergoing laparoscopic cholecystectomy, under general anesthesia, were randomly allocated in two groups. The first group received intravenous lidocaine infusion during the procedure until one hour postoperatively; meanwhile the second group received intravenous saline for the same period of time. The intervention was double-blind. In the postoperative period, both groups received dipyrone and morphine PCA. Pain was assessed by Visual Numeric Scale (VNS) at rest and when coughing at 1st, 2nd, 4th, 12th e 24th hour after the end of the surgery. Blood samples for cytokines measurement were taken at the end of procedure and 24 hours later. The total morphine PCA demand, the time for the first flatus and the length of hospital stay were also recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years and
* physical status according to the American Society of Anesthesiologists (ASA) I and II

Exclusion Criteria:

* patients older than 75 years,
* patients with heart disease,
* patients with history of:

  * kidney failure,
  * liver failure,
  * psychiatric disorder,
  * chronic use of opioids or medications that could cause induction of liver enzymes (anticonvulsants).
* the presentation of adverse effects during the intervention or postoperative complications, and the conversion to open surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome was pain intensity as assessed by visual analogical scale (VAS) scores | 24 hours
  The primary endpoint was the effect of lidocaine on postoperative pain within the first 24 hours. Three interns who participante of the study applied VNS to measure the intensity of pain at rest and when coughing 1, 2, 4, 12 and 24 hours after surgery.

SECONDARY OUTCOMES:
The secondary outcome was measure of citokynes IL-1 levels | 24 hours.
  A blood sample was collected by the author or by the anesthetist of the procedure to measure IL-1, IL-6, IL-10, TNF α and IFN γ levels immediately at the end of the surgery and 24 hours after. The difference of these markers between the two groups also featured secondary outcome. The samples were centrifuged and the serum was separated in Eppendorfs and then frozen at - 70 Celsius degrees, for posterior simultaneous analysis. The biochemical responsible for this analysis also did not have contact with the group to which participants belonged.
The secondary outcome was measure of citokynes IL-6 levels | 24 hours
  The primary endpoint was the effect of lidocaine on postoperative pain within the first 24 hours. Three interns who participante of the study applied VNS to measure the intensity of pain at rest and when coughing 1, 2, 4, 12 and 24 hours after surgery.
The secondary outcome was measure of citokynes IL-10 levels | 24 hours
  The primary endpoint was the effect of lidocaine on postoperative pain within the first 24 hours. Three interns who participante of the study applied VNS to measure the intensity of pain at rest and when coughing 1, 2, 4, 12 and 24 hours after surgery.
The secondary outcome was measure of citokynes TNF levels | 24 hours
  The primary endpoint was the effect of lidocaine on postoperative pain within the first 24 hours. Three interns who participante of the study applied VNS to measure the intensity of pain at rest and when coughing 1, 2, 4, 12 and 24 hours after surgery.
The secondary outcome was measure of citokynes IFN γ levels | 24 hours
  The primary endpoint was the effect of lidocaine on postoperative pain within the first 24 hours. Three interns who participante of the study applied VNS to measure the intensity of pain at rest and when coughing 1, 2, 4, 12 and 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Juliano Ferreira, PhD, Principal Investigator — Federal University of Santa Catarina